CLINICAL TRIAL: NCT03462641
Title: Modulation of GABA-A Receptors and Axial Motor Impairments in Parkinson Disease-Flumazenil Arm
Brief Title: Modulation of GABA-A Receptors in Parkinson Disease-Flumazenil Arm
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Nicolaas Bohnen, MD, PhD, Professor of Radiology and Neurology, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: HUM00130361; R01NS099535 (NIH)
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease
Keywords: Gait; Balance; Flumazenil; PET Imaging; MRI; Mobility; Intravenous
MeSH Terms: conditions — Parkinson Disease | interventions — Flumazenil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence A - (Flumazenil at Visit 1) (Experimental): A detailed 90 minute clinical assessment was conducted before and after treatment administration for each visit. Flumazenil 1mg in 10cc normal saline was given intravenously (iv) over 5-10 minutes on the first visit as treatment. 10 cc of normal saline placebo was given intravenously (iv) over 5-10 minutes on the second visit as treatment.
  Interventions: Drug: Flumazenil; Drug: Placebo
- Sequence B - (Placebo at Visit 1) (Experimental): A detailed 90 minute clinical assessment was conducted before and after treatment administration for each visit. 10 cc of normal saline placebo was given intravenously (iv) over 5-10 minutes on the first visit as treatment. Flumazenil 1mg in 10cc normal saline was given intravenously (iv) over 5-10 minutes on the second visit as treatment.
  Interventions: Drug: Flumazenil; Drug: Placebo

INTERVENTIONS:
Drug: Flumazenil — 1mg in 10cc normal saline
Drug: Placebo — 10 cc normal saline

SUMMARY:
This arm is a positron emission tomography (PET) biomechanistic GABA-A receptor target engagement study that includes detailed clinical and motor assessments before and after the i.v. administration of 1 mg flumazenil or placebo in Parkinson disease subjects. Each subject will receive 1mg flumazenil or placebo at two visits.

DETAILED DESCRIPTION:
This biomechanistic GABA-A receptor target engagement study includes clinical and motor assessments before and at various time points up to approximately 90 minutes after the i.v. administration of 1 mg flumazenil and placebo in Parkinson disease subjects. Thirty Parkinson disease subjects with disease severity (Hoehn and Yahr) stages 2-4 will be recruited. Baseline [11C]FMZ and vesicular monoamine transporter type 2 (VMAT2) [11C]DTBZ brain PET imaging will be performed prior to drug administration to assess for GABA-A receptor availability and the integrity of nigrostriatal dopaminergic nerve terminals, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Parkinson's disease (PD): PD diagnosis will follow the UK Parkinson's Disease Society Brain Bank Research Center (UKPDSBRC) clinical diagnostic criteria for PD.
2. Hoehn and Yahr stages 2-4
3. Absence of dementia confirmed by cognitive testing.
4. Abnormal 11C-Dihydrotetrabenazine ([11C]-DTBZ) PET study to demonstrate nigrostriatal dopaminergic denervation.

Exclusion Criteria:

1. PD with Dementia (PDD) or dementia with Lewy bodies (DLB).
2. Other disorders which may resemble PD, such as vascular dementia, normal pressure hydrocephalus, multiple system atrophy, corticobasal ganglionic degeneration, or toxic causes of parkinsonism. Prototypical cases have distinctive clinical profiles, like early and severe dysautonomia or appendicular apraxia, which may differentiate them from idiopathic PD. The use of the UKPDSBRC clinical diagnostic criteria for PD will mitigate the inclusion of subjects with atypical parkinsonism.
3. Subjects on benzodiazepine, GABA-ergic medications (baclofen, tizanidine), neuroleptic, anticholinergic (trihexyphenidyl, benztropine), or cholinesterase inhibitor drugs.
4. Evidence of a mass lesion on structural brain imaging (MRI).
5. Participants in whom MRI is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, chest, or cochlear implant.
6. Severe claustrophobia precluding MR or PET imaging.
7. Subjects limited by participation in research procedures involving ionizing radiation.
8. Pregnancy (urine or serum pregnancy test within 48 hours of each PET session) or breastfeeding.
9. History of seizures
10. Significant anxiety or history of panic disorder.
11. History of recent suicide attempt or overdose of tricyclic antidepressants or other medications
12. Any other medical history determined by investigators to preclude safe participation.
13. Allergy to flumazenil
14. Significant liver disease
15. History of alcohol or other substance abuse within past two years.
16. History of regular benzodiazepine use within past year

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas I Bohnen, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Functional Neuroimaging, Cognitive and Mobility Laboratory, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 36 people who consented, six were not actually randomized. One participant passed away for reasons unrelated to the study prior to assignment. One participant failed to complete the required dopaminergic PET scan. Two participants failed to show dopaminergic denervation on their PET scan, which was one of the exclusion criteria. Two participants withdrew prior to screening.
Period: Visit 1
Arm/Group | Sequence A - (Flumazenil at Visit 1) | Sequence B - (Placebo at Visit 1)
Started | 19 | 11
Actually Received Drug or Placebo | 18 | 11
Completed | 18 | 11
Not Completed | 1 | 0
Not completed — Failed to complete dopaminergic PET scan | 1 | 0
Period: Visit 2
Arm/Group | Sequence A - (Flumazenil at Visit 1) | Sequence B - (Placebo at Visit 1)
Started | 18 | 11
Actually Received Drug or Placebo | 18 | 10
Completed | 18 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: This is a per protocol analysis. Only the 28 participants that actually completed the entire study are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A - (Flumazenil at Visit 1) | Sequence B - (Placebo at Visit 1) | Total
Number analyzed (Participants) | 18 | 10 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.61 (5.85) | 69.5 (7.20) | 68.93 (6.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 13 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 10 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 9 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 10 | 28
Postural Instability and Gait Disorder score [Mean (Standard Deviation); unit: units on a scale] — Postural Instability and Gait Disorder (PIGD) score is a subscale score of Movement Disordered Society Sponsored Revision of the Unified Parkinsons Disease Rating Scale (MDS-UPDRS) scale.
  It is computed as a sum of following MDS-UPDRS items:
  3.10 Gait
  3.11 Freezing of gait
  3.12 Postural stability
  3.13 Posture
  Minimal possible score is 0, maximal possible score is 16. Higher scores indicate greater severity of PIGD symptoms (worse outcome).
  units on a scale | 5.64 (2.75) | 5.4 (2.28) | 5.55 (2.55)
Thalamic FMZ PET [Mean (Standard Deviation); unit: Parametric DVR] — Thalamic flumazenil (FMZ) binding was computed by averaging the dynamic resliced FMZ PET image across the 70 minute PET scanning session, and then normalizing the resulting values by the average value of the ventral pons reference region. Regional distribution volume ratio (DVR) were then extracted by taking the mean of voxels within each brain region and dividing it by the number of voxels in that brain region. Lastly, regional DVR were bilaterally averaged for this analysis, since we had no a-priori hypothesis about differences in hemispheric involvement for this analysis.
  Parametric DVR | 3.10 (0.24) | 3.14 (0.30) | 3.11 (0.26)

OUTCOME MEASURES:

1. Primary Outcome: Postural Instability and Gait Disorder (PIGD) Score
Description: Postural Instability and Gait Disorder (PIGD) score is a subscale score of MDS-UPDRS scale.
  It is computed as a sum of following MDS-UPDRS items:
  3.10 Gait
  3.11 Freezing of gait
  3.12 Postural stability
  3.13 Posture
  Minimal possible score is 0, maximal possible score is 16. Higher scores indicate greater severity of PIGD symptoms (worse outcome).
Time Frame: up to 3 hours (including pre and post infusion motor evaluation)
Population: MDS-UPDRS PIGD scores for the same set of 28 participants, recorded before and after treatment (placebo or flumazenil) administration.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: MDS-UPDRS PIGD score before treatment administration on the day when placebo was given.
- Flumazenil: MDS-UPDRS PIGD score before treatment administration on the day when flumazenil was given.
Arm/Group | Placebo | Flumazenil
Number analyzed (Participants) | 28 | 28
score on a scale
  Before Infusion | 4.625 (2.36) | 4.625 (2.34)
  After Infusion | 4.23 (2.15) | 4.09 (2.00)
Statistical Analysis 1: Comparison: Flumazenil; Null hypothesis was no difference in PIGD score within participants before and after flumazenil infusion; Test type: Superiority; p = 0.0407, Paired-Sample Two-Tailed T-Test — Alpha was set to 0.05; t-value = -2.15, Standard Deviation 1.32
Statistical Analysis 2: Comparison: Placebo vs Flumazenil; Null hypothesis is that there is no significant interaction between drug and time of administration (pre vs. post infusion); Test type: Other; p = 0.103, Repeated Measures ANCOVA — P value is given for the Drug*Time term, which represents interaction between time relative to administration (before infusion vs after infusion) and treatment administered (placebo vs flumazenil). Alpha was set to 0.05; F-value = 2.861

2. Primary Outcome: PIGD Score Change
Description: Difference in PIGD score from pre-infusion to post-infusion. Only observations where PIGD score change is less than 0 (decrease) are retained, as the hypothesis we are interested is whether the effect magnitude of flumazenil on PIGD score depends on baseline GABA-A receptor binding as assesed by FMZ PET.
Time Frame: up to 3 hours (including pre and post infusion motor evaluation)
Population: A subset of participants assigned to each sequence which showed a decrease in PIGD score from pre-infusion to post-infusion for placebo or flumazenil treatment. A total of 12 participants are included in this analysis, with some of them showing response in both placebo and flumazenil condition and others in one of the two.
Measure: Mean (Standard Deviation); unit: Change in PIGD Score
Groups:
- Placebo Responders: A subset of participants that showed a decreased PIGD score in response to placebo treatment.
- Flumazenil Responders: A subset of participants that showed a decreased PIGD score in response to flumazenil treatment.
Arm/Group | Placebo Responders | Flumazenil Responders
Number analyzed (Participants) | 8 | 6
Change in PIGD Score | -1.375 (0.5175492) | -2.500 (1.5165751)
Statistical Analysis 1: Comparison: Placebo Responders; A pair of maximum likelihood mixed linear models were estimated. The first was a random intercept model that merely accounted for individual differences in PIGD score before infusion. The second was an interaction model, that added an interaction term between baseline FMZ PET binding and PIGD score change from pre to post infusion. The interaction model was compared against the random intercept model to determine significance of the interaction using likelihood ratio goodness of fit test; Test type: Other; p = 0.00000029, Mixed Models Analysis — P value presented is for model comparison between interaction model and random intercept model; Standardized β Coefficient = 0.60, 95% CI 2-sided [0.13 to 1.07]

ADVERSE EVENTS:
Time Frame: up to 3 hours (including pre and post infusion motor evaluation)
Groups:
- Placebo Treatment: 10 cc of normal saline placebo was given intravenously (iv) over 5-10 minutes. A detailed 90 minute clinical assessment was conducted before and after treatment administration for each visit.
- Flumazenil Treatment: Flumazenil 1mg in 10cc normal saline was given intravenously (iv) over 5-10 minutes. 10 cc of normal saline placebo was given intravenously (iv) over 5-10 minutes. A detailed 90 minute clinical assessment was conducted before and after treatment administration for each visit.
Arm/Group | Placebo Treatment | Flumazenil Treatment
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28

LIMITATIONS AND CAVEATS:
Our participants were predominantly male, which is often the case with Parkinson's disease (PD) patient population since PD is known to affect males at a greater rate. This means that our findings may not generalize as well to population of female PD patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03462641/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT03462641/SAP_001.pdf